CLINICAL TRIAL: NCT04344743
Title: Cryoballoon Ablation Without Use of Contrast Dye for the Treatment of Paroxysmal Atrial Fibrillation
Brief Title: Balloon Cryoablation Without Contrast
Acronym: CRY-OUT-CAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medicover Hospital (Other)
Collaborators: National Institute of Cardiology, Warsaw, Poland (Other)
Responsible Party: Principal Investigator, Pawel Derejko, Head of Cardiology Department, Medicover Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1_2020
Record Dates: First submitted 2020-04-05; First posted 2020-04-14 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Cryoballoon ablation without contrast (Experimental): Cryoballoon ablation without contrast
  Interventions: Device: Cryoballoon ablation without contrast

INTERVENTIONS:
Device: Cryoballoon ablation without contrast — Cryoballoon ablation without contrast

SUMMARY:
Pulmonary vein isolation using cryoballoon ablation is well established method for the treatment of atrial fibrillation. As a rule, cryoenergy delivery is preceded by documenting the full vein occlusion. It is assessed by venography, performed by injecting contrast through the inner lumen of the balloon catheter after the vein is blocked with a balloon. Achieving full vein occlusion in certain situations can be challenging and may require multiple attempts, which may expose the patient to increased doses of contrast and radiation.. At the same time, the purpose of ablation is an electrical isolation of pulmonary veins.

Experts postulate ablation in the antrum and the so-called "proximal-seal technique", which in some cases may require to start cryoapplication before the vein is fully sealed. This approach minimizes the risk of the pulmonary vein stenosis, damage to structures immediately adjacent to the atrium and phrenic nerve palsy. In addition, in many cases the displacement of the balloon after several dozen seconds of cryoapplication, usually by pulling it, causes full sealing of the vein, contributes to further lowering the temperature and leads to full electrical isolation of the vein, which is the aims of ablation.

All the above-mentioned facts indicate that demonstrating full vein occlusion using angiography before the initiation of cryoenergy application is of limited value. Moreover, there are a number of parameters related to cryoballoon ablation that indicate acute and long term vein isolation.

Taking into account the arguments presented above, it seems that it is possible to perform an effective and safe isolation of the pulmonary veins using the cryoballoon ablation technique without confirmation by venography that PV is occluded. Along with dissemination of the method, such attempts are and will be made by some operators. Therefore, a systematic approach to this issue is important. It should define the conditions that should be met in order for the procedure in the proposed modification to be implemented effectively and safely. In addition, a protocol of ablation for this modification is required.

DETAILED DESCRIPTION:
Pulmonary vein isolation using cryoballoon ablation is well established method for the treatment of atrial fibrillation. As a rule, cryoenergy delivery is preceded by documenting the full vein occlusion. It is assessed by venography, performed by injecting contrast through the inner lumen of the balloon catheter after the vein is blocked with a balloon. Achieving full vein occlusion in certain situations can be challenging and may require multiple attempts, which may expose the patient to increased doses of contrast and radiation.. At the same time, the purpose of ablation is an electrical isolation of pulmonary veins.

Experts postulate ablation in the antrum and the so-called "proximal-seal technique", which in some cases may require to start cryoapplication before the vein is fully sealed. This approach minimizes the risk of the pulmonary vein stenosis, damage to structures immediately adjacent to the atrium and phrenic nerve palsy. In addition, in many cases the displacement of the balloon after several dozen seconds of cryoapplication, usually by pulling it, causes full sealing of the vein, contributes to further lowering the temperature and leads to full electrical isolation of the vein, which is the aims of ablation.

All the above-mentioned facts indicate that demonstrating full vein occlusion using angiography before the initiation of cryoenergy application is of limited value. Moreover, there are a number of parameters related to cryoballoon ablation that indicate acute and long term vein isolation.

Taking into account the arguments presented above, it seems that it is possible to perform an effective and safe isolation of the pulmonary veins using the cryoballoon ablation technique without confirmation by venography that PV is occluded. Along with dissemination of the method, such attempts are and will be made by some operators. Therefore, a systematic approach to this issue is important. It should define the conditions that should be met in order for the procedure in the proposed modification to be implemented effectively and safely. In addition, a protocol of ablation for this modification is required.

Course of ablation. All ablations will be performed using Medtronic Arctic Front Advance catheter system as well as future generations of Medtronic cryoballoon catheter systems.

Initially the cryoenergy will be delivered without previous venography confirming full vein occlusion. Then, in case of vein isolation failure after 5 minutes of cryoenergy delivery, further attempts to isolate the vein will be preceded by venography.

Statistical analysis. The assumed sample size (N = 50 patients/ 200 veins) will allow to estimate the number and percentage of pulmonary veins that will be isolated without the use of contrast.

The statistical analysis will use standard descriptive statistics tools: frequency tables for categorical variables; extreme values, mean value and standard deviation for normal distributed variables; and extreme values and quartiles for non-normal distributed variables.

Parameters assessed during the procedure:

Concerning a single energy cryoapplication

1. Possibility of registration (occurrence vs. non-occurrence) of pulmonary vein potentials before the cryoapplication, and after the occlusion of the vein by the balloon.
2. Time to vein isolation
3. Cryoenergy application time / freezing time
4. The minimum temperature obtained during cryoapplication
5. Time to obtain temperature - 30 ° C and - 40 ° C
6. Temperature after 30, 60 and 90 seconds from the beginning of cryoenergy application
7. Cryoballoon heating time from -30 C to +15 C Concerning the isolation of a single vein
8. Total time to complete isolation of a vein
9. The number of cryoenergy applications
10. Total time of cryoenergy application per vein

    Concerning the entire procedure:
11. Total cryoenergy application time per procedure / patient
12. The total amount of contrast
13. Radiation dose
14. Time of radiation
15. Left atrial dwelling time
16. Duration of the procedure (from puncture of the vein to sheaths removal)

Termination of cryoenergy delivery:

1. If temperature does not reach - 30 ° C after 60 seconds of cryoenergy application (inefficient application).
2. If vein isolation does not occur after 90 seconds of cryoenergy application (inefficient application).
3. If temperature after 30 seconds of cryoapplication falls lower than - 50° C (unsafe application).
4. When temperature reaches - 55° C (unsafe application).
5. If phrenic nerve injury occurs or if symptoms suggesting its imminent occurrence are noticed (unsafe application).
6. If the operator considers that the application is ineffective or performed too distally (inefficient or unsafe application).

Effective cryoenergy applications will be terminated 120 seconds after vein isolation.

Veins with no recordable pulmonary vein potentials - The above-mentioned veins will be isolated - 1 application 240 seconds. Applications will be considered effective if the minimum temperature achieved will be less than 35C and the stimulation performed from the vein after application will be ineffective.

Supplemental cryoapplications. Supplemental cryoenergy applications will not be delivered after successful isolation of the vein

Vein isolation assessment. Pulmonary vein isolation will be assessed by demonstrating entrance and exit block

Phrenic nerve function monitoring. In order to prevent PN injury/ palsy the balloon will be inflated outside PV ostia and maintained as antrally as possible during vein isolation. For phrenic nerve function monitoring pacing of the nerve during right pulmonary vein isolation will be performed. Additionally, intermittent fluoroscopy during pacing will be used for monitoring diaphragmatic motion. The ablation will be stopped at the first sign of imminent phrenic nerve injury.

Complications assessed. Transient phrenic nerve injury or palsy (resolving until discharge after index procedure) is considered a minor complication. Death, stroke, tamponade, arteriovenous fistula or pseudoaneurysm, persistent (resolving during follow up) or permanent (if not resolved at end of follow up, but >12 months) phrenic nerve palsy, bleeding with a decrease in haemoglobin of at least 2 g / dl or any other state requiring prolongation of hospitalization are considered major complications.

The duration of the project and follow-up. The study is expected to last two years. Approximately 50 patients will be enrolled, with one year follow-up. All patients will have follow-up visits in an out-patient clinic at least 3 and 12 months post PVI. Additionally at 6 weeks, 6 and 9 months post ablation telephone follow-up will be conducted by the study coordinator using standardized questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients with paroxysmal AF - episodes lasting up to 7 days or cardioverted before this time
* At least 4 AF attacks in the last 12 months
* Informed consent for participation in the study
* Age > 18 and < 70 years
* Left atrium diameter (PLAX) < 4,5 cm and left atrial area < = 30 cm2
* Left ventricle ejection fraction > 45%
* Four separate veins visualised in computed tomography prior to the ablation

Exclusion Criteria:

* Withdrawal of consent for the procedure
* Documented typical atrial flutter prior to the ablation
* Thrombus in left atrium
* GFR < 60 ml/min
* Pregnancy
* Common trunk of left or right pulmonary veins documented on computed tomography (preferred) or by means of other imaging methods
* Other conditions that preclude AF ablation including: infection, uncontrolled hyperthyroidism, significant anaemia and thrombocytopenia, acute cardiac / internist / surgical conditions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-08-13 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Isolation of a pulmonary vein without the use of contrast and within the scheduled timeframe | Through study completion, an average of 2 years
  Acute result will be assessed. Vein isolation assessment will be done using a diagnostic circular catheter (Achieve, Medtronic), by demonstrating entrance and exit block

SECONDARY OUTCOMES:
Percentage of patients in whom isolation of all pulmonary veins will be achieved without the use of contrast | Through study completion, an average of 2 years
Percentage of patients with stable sinus rhythm, without atrial fibrillation episodes during follow-up | During one year follow-up
The amount of contrast dye used | Through study completion, an average of 2 years
X-ray time exposure | Through study completion, an average of 2 years
Radiation dose | Through study completion, an average of 2 years
Left atrial dwelling time | Through study completion, an average of 2 years
Number of complications assessed | Through study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Pawel Derejko, MD, PhD, Principal Investigator — Medicover Hospital, Warsaw, Poland
Locations (2):
- Poland (2):
  - Medicover Hospital, Warsaw
  - National Institute of Cardiology, Warsaw

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables,figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.
  For individual participant data meta-analysis